CLINICAL TRIAL: NCT07280117
Title: Magnesium-based Bioresorbable Pins for Membrane Fixation in Case of Sinus Floor Elevation (SFE): a Prospective Case Series
Brief Title: Magnesium-based Bioresorbable Pins for Membrane Fixation
Status: Not yet recruiting | Type: Observational
Sponsor: Valentin Herber (Other)
Responsible Party: Sponsor-Investigator, Valentin Herber, Dr.med.dent., University of Basel
Organization: University of Basel (Other)
Other Study IDs: 2025-01789
Record Dates: First submitted 2025-12-01; First posted 2025-12-12 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-11

CONDITIONS: Sinus Floor Augmentation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

SUMMARY:
The goal of this research project is to assess the clinical performance and degradation of bioresorbable Mg- based pins for membrane fixation in patients with sinus floor elevation.

ELIGIBILITY:
Inclusion Criteria:

* Healthy patients in the aged > 21 years.
* fully or partially edentulous with unilaterally or bilaterally missing upper premolars or molars and an insufficient residual bone height to guarantee primary stability of implants; and requiring a staged approach of SFE and implant surgery
* Subject has been informed and signed the informed consent

Exclusion Criteria:

* Smoking more than 9 cigarettes per day
* Irradiation in the maxilla-facial region,
* A known metabolic skeletal disease (such as osteomalacia, osteoporosis or osteogenesis imperfecta) or medications that can affect the bone structure
* Allergies / intolerances to the materials
* Known malignancy
* Epilepsy or anamnestic evidence of recurrent falls
* Pregnancy (as contraindicated for CBCT imaging that is routinely performed)
* Manifest hepato-renal disease
* Inability or unwillingness to give informed consent.

Min Age: 21 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patient requiring a staged approach SFE
Sampling Method: Non-Probability Sample
Enrollment: 12 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2027-03-01 (Estimated); Study Completion 2028-08-01 (Estimated)

PRIMARY OUTCOMES:
Visually successful fixation of the membrane: | During SFE

SECONDARY OUTCOMES:
Material degradation of the Mg pins | after 6 months